CLINICAL TRIAL: NCT03814993
Title: Multicenter Observational Study to Determine the Long-term Tolerability and Analgesic Effectiveness of Oral Tapentadol in Patients Suffering From Severe Pain Syndromes, Refractory to Other Strong Opioids.
Brief Title: taPentadol cLinical prAcTice IN belgiUM
Acronym: PLATINUM
Status: Completed | Type: Observational
Sponsor: Dafne Balemans (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor-Investigator, Dafne Balemans, Clinical Trial Center UZA, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Other Study IDs: PLATINUM
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Severe Pain Syndromes
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Multicenter observational study to determine the long-term tolerability and analgesic effectiveness of oral tapentadol in patients suffering from severe pain syndromes, refractory to other strong opioids.

DETAILED DESCRIPTION:
Tapentadol, a centrally acting analgesic. It is indicated in Europe "for the relief of moderate to severe acute pain in adults, which can be adequately managed only with opioid analgesics" (IR formulation/oral solution) and "for the management of severe chronic pain in adults, which can be adequately managed only with opioid analgesics" (SR formulation). Tapentadol is reimbursed in Belgium since May 1, 2018. The reimbursement was obtained through an article 81 procedure (Chapter IV) which means that the reimbursement is currently restricted to the time frame of the contract and that during that period certain questions and uncertainties regarding the use of tapentadol in a Belgian setting need to be answered. In order to answer the questions raised by the Belgian Healthcare authorities, this study will be performed evaluating the application of oral tapentadol in routine clinical practice in Belgium. The study is conceived as a nation-wide multicentre prospective non-interventional trial. The primary endpoint and secondary endpoints of this study are guided by the questions that need to be answered during the course of the contract reimbursement, as established by the Belgian health authorities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be capable of giving their informed consent;
* Males and females, 18 years and older;
* Patients suffering from severe pain;
* Pain symptoms refractory to strong opioids (in previous treatment);

  * Due to side effects
  * Due to insufficient analgesic effectiveness
  * Due to opioid induced hyperalgesia.

Exclusion Criteria:

* Severe renal and/or hepatic insufficiency;
* Known and/or strong suspicion of allergy to tapentadol;
* Previous treatment with tapentadol;
* Presence of any condition for which tapentadol is contraindicated as per its approved labelling information in Belgium;
* The patient has no access to a mobile phone and web browser. During the study, an online system is used to receive messages (SMS and e-mail) for the completing of the online assessments (through web browser).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from severe pain that did not respond to previous treatment with strong opioids (either due to (1) insufficient analgesic effectiveness, (2) intolerable side effects from previous opioid treatment or (3) opioid induced hyperalgesia)
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Difference in occurrence of gastrointestinal side effects (nausea, vomiting and constipation) between baseline and week 15 | baseline - week 15
  Differences in occurence of the PRO-CTCAE items: Nausea, vomiting and constipation

SECONDARY OUTCOMES:
Difference in frequency, severity and interference of selected side effects (dizziness, fatigue, itching, headache, dry mouth, nausea, vomiting, constipation) from baseline to week 52 | baseline - week 52
  Difference in frequency, severity and interference of selected PRO-CTCAE items
Change From Baseline in Pain Scores on the Numeric Rating Scale baseline to different time points during long-term follow-up | baseline - week 52
  Reduction in pain intensity numeric rating scale (PI-NRS). Scale: 0 = no pain and 10 = worst possible pain
Change of health-related quality of life from baseline to different time points during long-term follow-up | baseline - week 52
  Change of healt-related quality of life measured by EQ-5D-5L (monthly evaluation)
Change of health-related quality of life from baseline to different time points during long-term follow-up | baseline - week 52
  Change of healt-related quality of life measured SF-36 (monthly evaluation)
Change of functional status of the patient from baseline to different time points during long-term follow-up | baseline - week 52
  Change of functional status measured by GPE-DV (monthly evaluation)
Change of functional status of the patient from baseline to different time points during long-term follow-up | baseline - week 52
  Change of functional status measured by impact pain on functioning (Interference-BPI)
Change of functional status of the patient from baseline to different time points during long-term follow-up | baseline - week 52
  Change of functional status measured by SF-36 (monthly evaluation)
The occurrence of tolerance during oral tapentadol treatment from baseline to different time points during long-term follow-up | baseline - week 52
  Occurence of tolerance by the use of MQS-III questionnaire (weekly or monthly)
The occurrence of tolerance during oral tapentadol treatment from baseline to different time points during long-term follow-up | baseline - week 52
  Occurence of tolerance by the use time-point of discontinuation of study drug
Drug conversion rates from other strong opioids to oral tapentadol from baseline to different time points during long-term follow-up | baseline - week 52
  By the use of MQS-III questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Guy Hans, Prof., Principal Investigator — University Hospital, Antwerp
Locations (11):
- Belgium (11):
  - AZ Monic, Antwerp
  - University Hospital Antwerp, Antwerp
  - Huisartspraktijk Van Peer, Boechout
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis Hasselt, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU Liège (Sart Tilman), Liège
  - Huisartspraktijk De Vaart, Mechelen
  - Grand Hôpital Charleroi, Montignies-sur-Sambre
  - AZ Turnhout, Turnhout